CLINICAL TRIAL: NCT00958620
Title: Shockwave Therapy of Chronic Achilles Tendinopathy. A Double-blind, Randomized Clinical Trial of Efficacy
Brief Title: Shockwave Therapy of Chronic Achilles Tendinopathy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Northern Orthopaedic Division, Denmark (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ON-07-001-RAS
Record Dates: First submitted 2009-08-12; First posted 2009-08-13 (Estimated); Last update posted 2015-05-28 (Estimated); Status verified 2015-05

CONDITIONS: Chronic Inflammatory Disorder
Keywords: Chronic Achilles Tendinopathy
MeSH Terms: interventions — Extracorporeal Shockwave Therapy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Active ESWT (Active Comparator)
  Interventions: Procedure: Shock Wave Therapy
- Sham ESWT (Sham Comparator)
  Interventions: Procedure: Shock Wave Therapy

INTERVENTIONS:
Procedure: Shock Wave Therapy — Extracorporal shock-wave therapy
  Other Names: Extracorporal shock-wave therapy

SUMMARY:
Chronic Achilles tendinopathy is a painful condition with frequently unsatisfactory results of conservative treatment. Extracorporal Shock Wave Therapy (ESWT) has been introduced in the management of various soft tissue conditions. The objective of the study was to investigate the effect of supplementary ESWT versus placebo to conservative treatment of chronic Achilles tendinopathy.

DETAILED DESCRIPTION:
Chronic Achilles tendinopathy is a common disability of the foot during walking and running. Avoiding of painful activities, correction of malalignment by arch support, stretching exercise and eccentric training combined with non-steroidal anti-inflammatory pain killers are the standard treatment regimen (Wilson 2005). However, evidence to support these modalities is sparse (McLauchlan 2001).

Extracorporal shock wave therapy (ESWT) originally used for treatment of renal stones became popular in the last decade for treatment of different soft tissue disorders including calcifying tendinopathy in the rotator cuff, humeral epicondylitis and plantar fasciitis (Haake 2001, Ogden 2001, Chung 2002, Gerdesmeyer 2003, Speed 2004). It is now worldwide employed and FDA-approved for the treatment of plantar fasciitis. However regarding both calcifying tendinopathy in the rotator cuff, humeral epicondylitis and plantar fasciitis the results are conflicting (Rompe 1996, Boddeker 2001, Hammer 2002, Schmitt 2002, Gross 2003, Haake 2003, Pleiner 2004, Chung 2005). A series of randomized studies on ESWT for soft tissue disorders have been reported (Rompe 1997, Krishek 1998, Loew 1999, Rompe 2001, Haake 2001, Hammer 2002, Schmitt 2002, Gerdesmeyer 2003, Gross 2003, Haake 2003, Pleiner 2004, Chung 2005, Costa 2005) only four reporting significant effect of ESWT (Rompe 1997, Krishek 1998, Loew 1999, Gerdesmeyer 2003), and only one randomised studies for chronic achilles tendinopathy (Costa 2005). Two uncontrolled (Perlick 2002, Lakshmanan 2003) and one controlled (Furia 2005) series introduce ESWT for chronic Achilles tendinopathy. The results of these papers are seriously conflicting. Some authors include training and others not. Since eccentric training has documented effect (Alfredson 2000) other conservative treatments should be introduced as a supplement.

We investigated in a double blind randomized trial the supplementary effect of ESWT to enhance recovery of Achilles tendinopathy. We investigated, firstly, the effect on AOFAS score and secondly the effect on pain.

ELIGIBILITY:
Inclusion criteria:

* Chronic Achilles Tendinopathy

Exclusion criteria:

* Recent surgery in area

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2004-10; Primary Completion 2005-01 (Actual); Study Completion 2005-06 (Actual)

PRIMARY OUTCOMES:
The American Orthopaedic Foot and Ankle Score (AOFAS score) | June 2005
Effect on pain | June 2005

CONTACTS AND LOCATIONS:
Overall Officials: Sten Rasmussen, MD, Principal Investigator — Orthopaedic Division, North Denmark Region, Aalborg University Hospital, Denmark